CLINICAL TRIAL: NCT01359436
Title: e- Ab Sensor-based Real-time Detection of Mutant EGFR in Clinical Specimens From Patients of Non-small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201007059R
Record Dates: First submitted 2011-05-23; First posted 2011-05-24 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-03

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electrosensing antibody probing system (e- Ab sensing) (Experimental)
  Interventions: Device: Electrosensing antibody probing system (e- Ab sensing)

INTERVENTIONS:
Device: Electrosensing antibody probing system (e- Ab sensing) — Electrosensing antibody probing system (e- Ab sensing), which was developed for the rapid and sensitive detection of hapten, proteins or viral antigen in medical samples, will be used for analyzing the interaction kinetics between mutation-specific anti-EGFR and its antigen mutant EGFR present in NSCLC. The system incorporates the use of engineered semiconductive antibodies or virus in vertical and lateral chip (eAbchip) or lateral flow through (eAbsignal) formats. In electrosensing antibody probing, semiconductive antibodies are bound as a suitable electrosensing probe which specifically and selectively binds mutant EGFR polypeptide target molecules in the test specimen.

SUMMARY:
The purpose of this study is to develop a real-time diagnostic technique with e- Ab sensor for specific EGFR mutation detection in clinical specimens of NSCLC patients, the investigators conduct a prospective clinical study. In comparison with results from direct sequencing of EGFR, the investigators evaluate the performance of e- Ab sensor, including reproducibility, sensitivity, specificity, and cross-reaction (such as detection of EGFR mutations other than L858R and DelL746-A750). The potential factors which may interfere with the results would be investigated. With such technique, the investigators can obtain EGFR mutation information of NSCLC patients in cost-saving and time-saving way and can offer more individualized treatment for the investigators patients.

DETAILED DESCRIPTION:
Epidermal growth factor receptor (EGFR) plays an important role in the development of non-small cell lung cancer (NSCLC). High EGFR mutation rate is found in certain population, including female, non-smoker, East Asian, and adenocarcinoma. Previous studies have shown that patients of NSCLC with mutant EGFR would have better survival, which was related to EGFR tyrosine kinase inhibitor treatment.1-2 IPASS study has shown that longer progression-free survival (PFS) under gefitinib treatment than that under carboplatin-paclitaxel, in patients with lung adenocarcinoma and clinical characteristics suggesting high EGFR mutation rate.3 However, only some EGFR mutations are associated with sensitivity to tyrosine kinase inhibitor treatment, especially deletion in exon 19 and L858R mutation in exon 21.4-5 Two recent phase III randomized clinical trials evaluated gefitinib treatment and chemotherapy in patients of advanced NSCLC with sensitive EGFR mutaions.6-7 In patients with advanced NSCLC and sensitive EGFR mutations, PFS under gefitinib was 9.2~10.8 months, longer than that under platinum-based chemotherapy. Therefore, to develop individualized treatment for patients with NSCLC, it is important to have EGFR mutation status at the time of diagnosis. Current techniques available for detection of EGFR mutation need direct sequencing of EGFR tyrosine kinase domains, which are costly and time-consuming. 8 For detection for specific EGFR mutations, mutation-specific monoclonal antibodies were developed to detect E746-A750 deletion in exon 19 and L858R in exon 21. In the pilot study, the immunohistochemistry (IHC) assay using mutation-specific antibodies showed a sensitivity of 92% and a specificity of 99%.9 Recent two studies examining the performance of the mutation-specific antibodies disclosed inconsistent sensitivity and specificity. In the study by Akhiko Kawahara et al, IHC assay of NSCLC tumor specimens with anti-delE746-A750 antibody showed a sensitivity of 79%, which was 83% by IHC assay with anti-L858R antibody.10 In the other study by Atsuko Kitamura et al, IHC assay with anti-delE746-A750 antibody showed high specificity but low sensitivity (99% and 40%, respectively). IHC assay with anti-L858R antibody also showed high specificity but low sensitivity (97% and 36%, respectively). The overall sensitivity and specificity of these two mutation-specific antibodies were 96% and 47%.11 The discrepancy between these two studies was currently unknown. Another study conducted in Memorial Sloan-Kettering Cancer Center showed the performance of these two mutation-specific antibodies would be affected by the cutoff of IHC score.12 For anti-L858R antibody, the sensitivity was 76%-95% and the positive predicted value was 99%-100%. For anti-delE746-A750 antibody, the sensitivity was 85%-67% and the positive predicted value was 99%-100%. It is unknown if the performance of these mutation-specific monoclonal antibodies could be enhanced with the use of automated quantitative system (AQUA). However, such techinique needs equipment and further cost, and couldn't offer immediate information about EGFR mutation to clinicians.

Electrosensing antibody probing system (e- Ab sensor), which was developed for the rapid and sensitive detection of hapten, proteins, or viral antigen in medical samples, will be used for analyzing the interaction kinetics between mutation specific anti-EGFR and its antigen (EGFR with E746-A750 deletion or L858R mutation) present in the specimens of patients with lung cancer. The system incorporates the use of engineered semiconducive antibodies or virus in vertical and lateral chip (eAbchip) or lateral flow through (eAbsignal) formats. In electrosensing antibody probing, semiconductive antibodies are bound as a suitable electrosensing probe, which specifically and selectively binds targeted molecules (i.e. specific mutant EGFR) in the test specimens. From assessment of the electric signature of semiconductive mutation-specific anti-EGFR antibodies, the eABprobe could offer sensitive detection and precise quantification of specific mutant EGFR.

To develop a real-time diagnostic technique with e- Ab sensor for specific EGFR mutation detection in clinical specimens of NSCLC patients, we conduct a prospective clinical study. In comparison with results from direct sequencing of EGFR, we evaluate the performance of e- Ab sensor, including reproducibility, sensitivity, specificity, and cross-reaction (such as detection of EGFR mutations other than L858R and DelL746-A750). The potential factors which may interfere with the results would be investigated. With such technique, we can obtain EGFR mutation information of NSCLC patients in cost-saving and time-saving way and can offer more individualized treatment for our patients.

ELIGIBILITY:
Inclusion Criteria:

Inclusion: Patients will be enrolled if they fulfill all of the following criteria

1. With indication for the following interventions:

   Thoracentesis Fine-needle aspiration and biopsy of primary tumor or metastases Bronchoalveolar lavage
2. With enough residual specimens for further study (Patients would be excluded if they have only limited amount of clinical specimens, which should all be sent for clinical analysis.)
3. Consent is obtained from the patient

Exclusion Criteria:

* Patients will be excluded if they couldn't sign the consent. Otherwise, no specific exclusion criteria were considered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The performance of e- Ab sensor | 1 day
  In comparison with results from direct sequencing of EGFR, we evaluate the performance of e- Ab sensor, including reproducibility, sensitivity, specificity, and cross-reaction (such as detection of EGFR mutations other than L858R and DelL746-A750)

CONTACTS AND LOCATIONS:
Overall Officials: Pan-Chyr Yang, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan